CLINICAL TRIAL: NCT06798246
Title: Hematoxylin-eosin Staining-based Tumor Microenvironment Subtype System Adjuvant Therapeutic Selection for Locally Advanced Upper Tract Urothelial Carcinoma After Radical Surgery：A Perspective Cohort Study
Brief Title: HEFTME System for Adjuvant Therapeutic Selection of Locally Advanced UTUC Postoperatively：A Perspective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Peking University Third Hospital (Other); Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Xuesong Li, Director of Department of Urology, Peking University First Hospital, Peking University First Hospital
Other Study IDs: TSU-04
Record Dates: First submitted 2024-12-08; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Upper Tract Urothelial Carcinoma
Keywords: HE-stained slides; Tumor microenvironment; Precise subtype; Adjuvant therapy
MeSH Terms: interventions — Drug Therapy; Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- D subtype: Participants were classified into four subtypes based on various combinations of TSR and sTIL scores: Depleted (D, TSR-low&sTIL-low)
  Interventions: Drug: Chemotherapy
- F subtype: Participants were classified into four subtypes based on various combinations of TSR and sTIL scores: Fibrotic (F, TSR-high&sTIL-low)
  Interventions: Drug: Chemotherapy combined with immunotherapy
- IE subtpye: Participants were classified into four subtypes based on various combinations of TSR and sTIL scores: Immune Enriched, Non-Fibrotic (IE, TSR-low&sTIL-high)
  Interventions: Drug: Immunotherapy
- IE/F subtype: Participants were classified into four subtypes based on various combinations of TSR and sTIL scores: Immune Enriched and Fibrotic (IE/F, TSR-high&sTIL-high)
  Interventions: Drug: ADC

INTERVENTIONS:
Drug: Chemotherapy — Gemicitabin and cisplatin
  Groups: D subtype
Drug: Immunotherapy — PD-1/PD-L1
  Groups: IE subtpye
Drug: ADC — ADC drug like RC48
  Groups: IE/F subtype
Drug: Chemotherapy combined with immunotherapy — Chemotherapy combined with immunotherapy
  Groups: F subtype

SUMMARY:
This multicenter, real-world study introduces a novel Hematoxylin-eosin staining(H&E)-based four tumor microenvironment (TME) system (HEFTME system) assisting in prognostic prediction and precise adjuvant treatment selection for laUTUC postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* pathological diagnose of UTUC;
* Met more than muscle-invasion stages(pT2+) or lymph nodes metastasis.

Exclusion Criteria:

* Patients with early-local stages (pTa/T1/Tis) without LNM+ and those with incomplete pathologic and prognostic information were excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced UTUC patients such as pathological diagnosed as UTUC with muscle-invasion stages or lymph nodes metastasis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
DFS | 1 year, 3 years and 5 years
  Disease-free survival include death and recurrence

SECONDARY OUTCOMES:
ORR | 3 month after the start of treatment until the end of treatment
  Response rate
OS | 1 year, 3 years and 5 years
  Overall survival
AE | 1-3 months after starting treatment
  adverse effects

IPD SHARING:
Plan to Share IPD: Yes
http://ai.yorktal.com
Supporting Information: Study Protocol